CLINICAL TRIAL: NCT06252688
Title: Conceptualisation of a Network Approach to Complete the Classification of Eating Disorders With the Aim of Better Personalising Their Management
Acronym: CASCADE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0261
Record Dates: First submitted 2023-11-17; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-09

CONDITIONS: Eating Disorders; Eating Disorder Binge
Keywords: Anorexia nervosa; Bulimia; Binge eating disorders; Neuropsychology; Neurocognitiond; Daily functioning
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Anorexia Nervosa; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): All participants performed the same evaluation: clinical and neuropsychological assessment.
  All of them are patients with an eating disorder.
  Interventions: Behavioral: Ambulatory cares in a day-hospital (Lapeyronie, Montpellier) specialized in the evaluation of eating disorders.

INTERVENTIONS:
Behavioral: Ambulatory cares in a day-hospital (Lapeyronie, Montpellier) specialized in the evaluation of eating disorders. — All patients assessed in the day-hospital will permormed the same evaluation :
  * Blood sampling
  * Calorimetry
  * Osteodensotometry
  * Psychiatric assement
  * Endocrinologic assessment
  * Dietetic assessment
  * Neuropsychological assessment
  * Self-questionnaires
  With the patient agreement, a biological collection will be constituted. The objective is the subsequent study of biological factors involved in eating disorders (in particular genetic factors)

SUMMARY:
Eating disorders (EDBs) are mental disorders with a great impact on the lives of individuals as well as a great cost imposed on society. The treatments currently available rely on different forms of psychotherapies with an unsatisfactory response rate as well as a considerable relapse rate . One of the reasons underlying the low success of available therapeutic modalities would be the heterogeneity of the clinical presentation of EDs, making their classification and the personalization of their treatment more difficult.The investigators hypothesize that a secondarily dimensional classification approach (respecting the categorical classification currently in use) of EDs based on the different dimensions disturbed in these disorders as well as in their comorbidities, would better represent their nosographic reality, which could provide patients with more personalized and potentially more effective care.

DETAILED DESCRIPTION:
Detailed Description:

The investigators will recruit a total of 840 patients with an eating disorder in the university hospital of Montpellier.

- Participation consists of a one-day visit with a multidisciplinary assessment. No action is specific to research except the biological collection for the constitution of a genetic bank. This is the usual management of patients with eating disorders addressed to our department.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an eating disorder according to DSM-V criteria
* Patient aged from 15 to 65 years
* Patient who performs the day-hospital evaluation
* Patient affiliated to a French social security system
* Patient able to understand the nature, the aim and the methodology of the study
* For minor one of the legal guardians gave his consent

Exclusion Criteria:

* Patient in an unstable somatic state (eg severe metabolic disorder making impossible or unreliable neuropsychological assessments)
* Patient's refusal to participate
* Patient protected by law (guardianship or curatorship)*
* Pregnant or nursing women. A dosage of βHCG will be performed to ensure the absence of pregnancy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2031-11-15 (Estimated); Study Completion 2031-11-15 (Estimated)

PRIMARY OUTCOMES:
Eating Disorders Inventory (EDI-2) | Baseline
  self-questionnaire of 91 items aimed at evaluating attitudes and behaviors related to food and allowing the identification of 11 dimensions: search for thinness, bulimia, body dissatisfaction, inefficiency, perfectionism, interpersonal distrust, interoceptive awareness, fear of maturity , asceticism, impulse control, social insecurity. The higher the subscore, the more severely impaired the dimension concerned is.
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline
  Self-reported version of the gold-standard clinical interview for ED assessing the intensity of eating symptoms over the last 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6 are thus obtained.

SECONDARY OUTCOMES:
Symptomatic dimensions of Eating Disorder Examination Questionnaire (EDEQ) | baseline
  Self-reported version of the gold-standard clinical interview for ED assessing the intensity of eating symptoms over the last 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6 are thus obtained.
Body Shape Questionnaire (BSAQ-34) | baseline
  self-questionnaire of 34 items assessing body dissatisfaction and in particular four dimensions: avoidance and social shame of body exposure, body dissatisfaction with the lower parts of the body, use of laxatives and vomiting to reduce body dissatisfaction, maladaptive cognitions and behaviors in order to control weight. The total score ranges from 0 to 204. A score below 80 indicates no excessive body concerns, a score between 80 and 100 indicates mild concerns, between 111 and 140 moderate concerns, and a score above 140 indicates significant concerns
Yale Food Addiction Scale (YFAS) | baseline
  35-item Likert-type self-questionnaire assessing the difficulty or not in controlling the quantity of food one eats over the past 12 months, using an 8-point scale from "never" to "all days ". This questionnaire assesses clinical distress based on the DSM-5 diagnostic criteria for substance use disorders. Presenting clinically significant suffering and at least 2 diagnostic criteria suggest a food addiction.
Sociocultural Attitudes Towards Appearance Scale (SATAQ-4) | baseline
  multidimensional self-questionnaire of 22 items rated from 1 (completely disagree) to 5 (completely agree) aimed at assessing the sociocultural influence of the media on appearance. It includes four subscales: pressures, information, internalization relating to athletes and general internalization. The higher the score, the stronger the influence.
Female drive for muscularity scale (FDMS) | baseline
  10-item self-questionnaire assessing the desire for muscularity in women. Each item is rated from 1 (never) to 6 (always). A high score indicates a significant search for musculature.
exercice and Eating disorders questionnaire (EED) | baseline
  self-questionnaire of 21 questions evaluating the different types of exercises (normal and pathological) carried out over the last 4 weeks. A high score suggests physical hyperactivity linked to food and body concerns.
Childhood Trauma Questionnaire (CTQ) | baseline
  28-item self-questionnaire that assesses past history of childhood abuse. 5 forms of mistreatment are assessed: physical abuse and sexual abuse, emotional abuse and emotional neglect, as well as physical neglect.
depression scale (PQ-9) | baseline
  self-assessment questionnaire measuring the severity of depression, composed of 9 items rated from 0 to 3. A total score varying from 0 to 27 is thus obtained. The higher the score, the more severe the depression.
The anxiety scale (GAD-7) | baseline
  self-questionnaire for assessing current anxious symptomatology consists of 7 items rated from 0 to 3. The total score ranges from 0 to 21. The recommended threshold for estimating generalized anxiety is 10.
The insomnia severity index (ISI) | baseline
  Sleep disorders are common in EDs. The ISI is a self-questionnaire of 5 items rated from 0 to 4 which makes it possible to assess the nature of insomnia, satisfaction with sleep, daily functioning and anxiety in relation to sleep disorders. A total score varying from 0 to 28 makes it possible to assess the severity of insomnia.
The disgust propensity and sensitivity scale (DPSS-R) | Baseline
  This scale of 10 items rated from 1 (never) to 5 (always) assesses sensitivity to disgust and is used to calibrate the level of exposure during treatment. The higher the score, the more sensitive the subjects are to the emotion of disgust.
The emotional regulation scale (DERS-F) | baseline
  This scale includes 36 items and aims to assess difficulties in regulating emotions through 6 dimensions: N (Non-acceptance): non-acceptance of one's emotional response, G (Goals): difficulties in adopting goal-oriented behaviors in a negative emotional context, I (Impulse): difficulties in controlling oneself in a negative emotional context, A (Awareness): lack of emotional awareness, S (Strategies): difficulties in implementing emotion regulation strategies in an emotional context negative, C (Clarity): difficulty identifying one's own emotions. The higher the score, the more difficulty the subject presents in regulating their emotions.
The Sheehan Global Functioning Scale (SDS) | baseline
  measures from 0 to 10, in self-assessment, the intensity of discomfort and handicap felt in three areas of professional, social and family functioning.
Detail and flexibility questionnaire (Dflex) | baseline
  24-item self-questionnaire measuring two aspects of neurocognitive functioning, rigidity (12 items) and lack of central coherence (12 items), as they manifest in a daily context. The two scores can vary from 12 to 72. The higher they are, the greater the perceived difficulties.
Rey's figure | baseline
  This is a test of copying and reproducing from memory a complex figure. The test draws on the subject's general intelligence abilities as well as their perceptual structuring skills. The purpose of the test in our study is to assess levels of central coherence (the ability to assess a situation as a whole rather than focusing on details).
d2 attention test | Baseline
  cancellation test where individuals must search for target items "d" with two dots among distractors across a series of 658 consecutively ordered items. Participants are instructed to cancel as many target symbols as possible by moving across the page in a manner similar to reading from left to right with a limit of 20 seconds per trial without interruption. The ratio between the number of omission errors (number of "d"s with two unmarked points) and the total number of items processed was the main variable considered in this study.
Wisconsin test (WCST-64) | Baseline
  This test explores executive functions using a set of 64 cards illustrated by the combination of three attributes: shape (cross, circle, triangle, star), color (yellow, red, blue, green) and number of figures (of 1 to 4). Four target cards are placed in front of the subject who must find a predetermined classification rule by trial and error. The results are expressed in number of categories completed, percentage of perseverative errors, number of trials necessary to complete the first category and learning capacity.
Delay discounting task (DDT) | Baseline
  This task evaluates decision-making abilities in a situation of projection into the future and makes it possible to suggest prognoses for development in TCA.
Mini International Neuropsychiatric Interview | Baseline
  MINI 5.0.0 allowing current and entire life diagnoses according to Axis-I of the DSM-5-TR
The relationship between BMI and the biological parameters of the blood test | Baseline
  The investigators want to study the link between the BMI and the alteration of the biological balance (ionogram, hetapic, liver function, hematogy corresponding to the standard biological assessment). (weight and height will be combined to report BMI in kg/m^2).
The relationship between disease duration and the biological parameters of the blood test | Baseline
  The investigators want to study the link between the disease duration and the alteration of the biological balance.
The relationship between BMI and calorimetry data | Baseline
  The investigators want to study the link between BMI and alteration of basal metabolism . (weight and height will be combined to report BMI in kg/m^2) Basal metabolims is the rate at which the body uses energy while at rest to maintain vital functions such as breathing and keeping warm (in Kcal per day)
The relationship between disease duration and calorimetry data | Baseline
  The investigators want to study the link between disease duration and alteration of basal metabolism.
  Basal metabolims is the rate at which the body uses energy while at rest to maintain vital functions such as breathing and keeping warm (in Kcal per day)
The relationship between BMI of TCA and bone densitometry data | Baseline
  The investigators want to study the link between BMI and Z score of bone demineralization. (weight and height will be combined to report BMI in kg/m^2) We aimed to asssess level of osteopenia compared to a reference population
The relationship between BMI and impedancemetry data | Baseline
  The investigators want to study the link between BMI and alterations in body composition (percentage of fat mass). (weight and height will be combined to report BMI in kg/m^2)
The relationship between disease duration and impedancemetry data | Baseline
  The investigators want to study the link between disease duration (in year) and alterations in body composition (percentage of fat mass).